CLINICAL TRIAL: NCT02906384
Title: Memory Preservation and Functional Brain Magnetic Resonance Imaging Changes With Conformal Avoidance of the Hippocampal Neural Stem-cell Compartment During Prophylactic Cranial Irradiation for Small Cell Lung Cancer Patients: A Prospective, Randomized Phase-II Study
Brief Title: Memory and MRI Changes With Hippocampus Avoidance Prophylactic Cranial Irradiation(HA-PCI) for Small Cell Lung Cancer(SCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-HA-PCI
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Small Cell Lung Cancer
Keywords: hippocampus avoidance; volumetric modulated arc therapy; functional MRI; hopkins Verbal Learning Test; prophylactic cranial irradiation
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- routine PCI (No Intervention): PTV:25Gy/10F. Radiation technique: VMAT.
- HA-PCI (Experimental): PTV 25Gy/10F. Hippocampus avoidance: decrease the dose to HAZ as the following criteria: Dmin<9Gy Dmax<16Gy.
  Radiation technique: VMAT.
  Interventions: Radiation: hippocampus avoidance

INTERVENTIONS:
Radiation: hippocampus avoidance — conformal avoidance of the hippocampal neural stem-cell compartment during prophylactic cranial irradiation
  Arms: HA-PCI

SUMMARY:
This is a prospective, randomized phase-II study observing the memory preservation and functional brain MRI changes with conformal avoidance of the hippocampal neural stem-cell compartment during prophylactic cranial irradiation for small cell lung cancer patients.

DETAILED DESCRIPTION:
Brain metastasis is rather high in small cell lung cancer patients. Prophylactic cranial irradiation(PCI) is the standardized treatment. However, cognitive dysfunction like memory damage is observed in quite a number of patients after brain irradiation, which may due to the hippocampus being irradiated. Thus, the investigators conduct the study by reducing the dose to the hippocampal neural stem-cell compartment (HAZ) during PCI.

Patient Population: Age: 18-65y; small cell lung cancer undergoing PCI; Eastern Cooperative Oncology Group (ECOG) score: 0-1.

The patients are randomized to 2 arms:

Arm Routine PCI: PTV(planning target volume) 25Gy/10F. Arm Hippocampus avoidance PCI(HA-PCI): PTV 25Gray(Gy)/10Fraction(F), HAZ Dmin<9Gy Dmax<16Gy).

Measurements: Hopkins verbal learning test(HVLT) and functional brain magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically conformed small cell lung cancer;
2. Complete response (CR)/partial response (PR) after chemo-radiotherapy;
3. ECOG (Eastern Cooperative Oncology Group) : 0-1;
4. No imaging evidence of brain metastasis before PCI;
5. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function);
6. Able to understand this study and have signed informed consent.

Exclusion Criteria:

1. Unable to receive MRI;
2. Medical history of central nervous system, cognitive or psychological diseases;
3. The expectation of life is less than 6 months;
4. Female in pregnancy or lactating;
5. The researchers consider the patient not appropriate to be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
memory preservation | 2 years
  responses to Hopkins Verbal Learning Test

SECONDARY OUTCOMES:
overall survival | 2 years
  Overall survival will be evaluated
hippocampus metastasis | 2 years
  hippocampus metastasis rate will be recorded
image changes of brain | 2 years
  changes of functional brain MRI will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, PHD, Principal Investigator — Zhejiang Cancer Hospital; Yue Kong, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No